CLINICAL TRIAL: NCT05539664
Title: A Prospective, Multi-center, Randomized, Controlled Clinical Trial to Evaluate the Effectiveness and Safety of Hydrogen-Oxygen Generator With Nebulizer for Adjuvant Treatment of 2019 Novel Coronavirus Pneumonia (COVID-19) Positive Patients
Brief Title: Hydrogen-Oxygen Generator With Nebulizer for Adjuvant Treatment of COVID-19 Positive Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMS-H-03-103
Record Dates: First submitted 2022-08-14; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-05

CONDITIONS: Covid19; Hydrogen-oxygen Gas; AMS-H-03
Keywords: Covid19; Hydrogen-oxygen Gas; AMS-H-03
MeSH Terms: conditions — COVID-19 | interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Intervention Model Description: The test group will use the investigational medical device Hydrogen-Oxygen Generator with Nebulizer (Shanghai Asclepius Meditec Co., Ltd.) + basic treatment (the investigator provides corresponding symptomatic support treatment based on the condition of the patients), and the control group will use the hospital routine oxygen supply equipment (wall oxygen or cylinder oxygen) + basic treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental Group (Experimental): The test group will use the investigational medical device Hydrogen-Oxygen Generator with Nebulizer (Shanghai Asclepius Meditec Co., Ltd.) + basic treatment (the investigator provides corresponding symptomatic support treatment based on the condition of the patients)
  Interventions: Device: Hydrogen-Oxygen Generator with Nebulizer, AMS-H-03
- Control Group (Active Comparator): The control group will use the hospital routine oxygen supply equipment (wall oxygen or cylinder oxygen) + basic treatment
  Interventions: Device: the hospital routine oxygen supply equipment (wall oxygen or cylinder oxygen)

INTERVENTIONS:
Device: Hydrogen-Oxygen Generator with Nebulizer, AMS-H-03 — The experimental group used the experimental medical device Hydrogen-Oxygen Generator with Nebulizer(Shanghai Asclepius Meditec Co., Ltd. ) The flow rate was 3L/min, and the cumulative treatment time was not less than 6 hours per day.
  Arms: experimental Group
Device: the hospital routine oxygen supply equipment (wall oxygen or cylinder oxygen) — the hospital routine oxygen supply equipment (wall oxygen or cylinder oxygen). The flow rate was 3L/min, and the cumulative treatment time was not less than 6 hours per day.
  Arms: Control Group

SUMMARY:
This is a prospective, multicenter, randomized, controlled, superiority clinical trial. It is expected that the test group would have better effectiveness than the control group in the primary evaluation indicator (time to negative viral nucleic acid detection from the start of study treatment). The test group will use the investigational medical device Hydrogen-Oxygen Generator with Nebulizer (Shanghai Asclepius Meditec Co., Ltd.) + basic treatment (the investigator provides corresponding symptomatic support treatment based on the condition of the patients), and the control group will use the hospital routine oxygen supply equipment (wall oxygen or cylinder oxygen) + basic treatment, to evaluate the effectiveness and safety of the investigational medical device Hydrogen-Oxygen Generator with Nebulizer for adjuvant treatment of COVID-19 patients.

DETAILED DESCRIPTION:
A total of 188 subjects who met the requirements of this study will be randomized into the test group or the control group in a 1:1 ratio to receive treatment, and the subjects will be observed and evaluated in the period from treatment after enrollment to discharge.

All enrolled subjects will receive treatment and visit, including screening visit (within 3 days before enrollment), randomization and treatment visit (Day 0), 1, 2, 3, 5, 7, 10, and discharge visit after treatment.

The primary effectiveness evaluation indicator (time to negative viral nucleic acid detection from the start of the study treatment), the secondary effectiveness evaluation indicators (viral nucleic acid negative conversion rate, imaging evaluation, inflammatory indicators such as CRP, IL-6, lymphocytes, clinical response rate at 7 days of treatment, recovery rate and recovery time of major symptoms, index oxygen saturation, and Ct value of nucleic acid detection), and safety evaluation indicators ( incidence of AE and SAE, incidence of device deficiencies) of the two groups will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged between 18 and 80 years old (inclusive).
* Diagnosed as general type of COVID-19 according to the criteria of Scheme for Diagnosis and Treatment of 2019 Novel Coronavirus Pneumonia (Trial Version 9).
* Subjects who are willing to participate and provided written informed consent form.

Exclusion Criteria:

* Diagnosed as mild, severe, critical or asymptomatic type of COVID-19.
* Subjects in the treatment or active stage of malignant tumor.
* Subjects who are intolerable to inhalation treatment.
* Subjects with mental disorders or cognitive impairment who are unable to provide consent.
* Subjects with any immunodeficiency requiring chronic treatment with any corticosteroid or other immunosuppressants.
* Complicate serious primary diseases such as heart, liver, kidney, and hematopoietic diseases; acute exacerbation phase of chronic obstructive pulmonary disease, or acute attack of bronchial asthma.
* Subjects who are using any non-expectorant antioxidant drug, including large doses of vitamin C and vitamin E.
* Subjects who are participating any other clinical study of any investigational drug or medical device.
* Pregnant or lactating women.
* Any other condition judged as inappropriate to participate in this study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to negative viral nucleic acid detection from the start of the study treatment. | through study completion, The average time from enrollment to two consecutive negative nucleic acid tests of respiratory specimens (sampling time interval of at least 24 hours) was approximately 7 days
  Time to negative viral nucleic acid detection is defined as two consecutive negative viral nucleic acid detections of respiratory specimens (samples will be taken at least 24 hours apart).

SECONDARY OUTCOMES:
Negative rate based on viral nucleic acid detection | The negative rate of viral nucleic acid detection from 3, 5, 7, 10 days after the treatment to discharge will be analyzed.
  Negative viral nucleic acid detection is defined as two consecutive negative nucleic acid detections of respiratory specimens (the sampling time interval will be at least 24 hours).
Imaging evalution indicators | Lung imaging changes were analyzed on the 3rd and 7th day after treatment.
  Significant lesion absorption >50%, lesion absorption degree of 10%-50%, lesion absorption degree of < 10%, and lesion progression compared with that at enrollment as showed in lung imaging.
CRP | The changes were compared with those on day 3, 5 and 7 before treatment.
  Inflammatory indicators such as CRP
Clinical effectiveness within 7 days | The clinical effective rate after 7 days of treatment will be used as the evaluation indiactor
  Clinically effective is defined as "cured" + "significant effective" + "effective". Clinical response rate = (total number of patients of "cured" + "significant effective" + "effective")/total number of subjects included in the analysis ×100%. It should be noted that in the actual situation, some clinical symptoms or signs may still be observed in the follow up after the end of treatment. If it is indicated that the above situation is resulted from the underlying disease, the investigator can also consider the patient to be clinically cured after comprehensive judgment based on the clinical data.
recovery rate and time to recovery of main symptoms | The patients will be followed up at 3, 5, 7, 10 days after the treatment and at discharge visit.
  It is defined as all major symptoms (fever, fatigue, cough, expectoration, chest tightness, chest pain, shortness of breath, and dyspnea) at enrollment had all disappeared or completely returned to normal at follow up.
Oxygen saturation | This will be evaluated at 3, 5, 7, and 10 days after the treatment and at discharge. The oxygen saturation will be measured at rest after stopping oxygen or hydrogen inhalation for 10 minutes.
  Oxygen saturation
Ct value in nucleic acid detection | This will be evaluated at1,2，3, 5, 7, and 10 days after the treatment and at discharge.
  Ct value in nucleic acid detection
IL-6 | The changes were compared with those on day 3, 5 and 7 before treatment.
  Inflammatory indicators such as IL-6
lymphocytes | The changes were compared with those on day 3, 5 and 7 before treatment.
  Inflammatory indicators such as lymphocytes

OTHER OUTCOMES:
AE/SAE percentage | through study completion, an average of 6 months
  AE/SAE percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Medical School of Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ksiazek TG, Erdman D, Goldsmith CS, Zaki SR, Peret T, Emery S, Tong S, Urbani C, Comer JA, Lim W, Rollin PE, Dowell SF, Ling AE, Humphrey CD, Shieh WJ, Guarner J, Paddock CD, Rota P, Fields B, DeRisi J, Yang JY, Cox N, Hughes JM, LeDuc JW, Bellini WJ, Anderson LJ; SARS Working Group. A novel coronavirus associated with severe acute respiratory syndrome. N Engl J Med. 2003 May 15;348(20):1953-66. doi: 10.1056/NEJMoa030781. Epub 2003 Apr 10. PMID 12690092
- [Background] Kuiken T, Fouchier RA, Schutten M, Rimmelzwaan GF, van Amerongen G, van Riel D, Laman JD, de Jong T, van Doornum G, Lim W, Ling AE, Chan PK, Tam JS, Zambon MC, Gopal R, Drosten C, van der Werf S, Escriou N, Manuguerra JC, Stohr K, Peiris JS, Osterhaus AD. Newly discovered coronavirus as the primary cause of severe acute respiratory syndrome. Lancet. 2003 Jul 26;362(9380):263-70. doi: 10.1016/S0140-6736(03)13967-0. PMID 12892955
- [Background] Drosten C, Gunther S, Preiser W, van der Werf S, Brodt HR, Becker S, Rabenau H, Panning M, Kolesnikova L, Fouchier RA, Berger A, Burguiere AM, Cinatl J, Eickmann M, Escriou N, Grywna K, Kramme S, Manuguerra JC, Muller S, Rickerts V, Sturmer M, Vieth S, Klenk HD, Osterhaus AD, Schmitz H, Doerr HW. Identification of a novel coronavirus in patients with severe acute respiratory syndrome. N Engl J Med. 2003 May 15;348(20):1967-76. doi: 10.1056/NEJMoa030747. Epub 2003 Apr 10. PMID 12690091
- [Background] de Groot RJ, Baker SC, Baric RS, Brown CS, Drosten C, Enjuanes L, Fouchier RA, Galiano M, Gorbalenya AE, Memish ZA, Perlman S, Poon LL, Snijder EJ, Stephens GM, Woo PC, Zaki AM, Zambon M, Ziebuhr J. Middle East respiratory syndrome coronavirus (MERS-CoV): announcement of the Coronavirus Study Group. J Virol. 2013 Jul;87(14):7790-2. doi: 10.1128/JVI.01244-13. Epub 2013 May 15. No abstract available. PMID 23678167
- [Background] Zaki AM, van Boheemen S, Bestebroer TM, Osterhaus AD, Fouchier RA. Isolation of a novel coronavirus from a man with pneumonia in Saudi Arabia. N Engl J Med. 2012 Nov 8;367(19):1814-20. doi: 10.1056/NEJMoa1211721. Epub 2012 Oct 17. PMID 23075143
- [Background] Zhou ZQ, Zhong CH, Su ZQ, Li XY, Chen Y, Chen XB, Tang CL, Zhou LQ, Li SY. Breathing Hydrogen-Oxygen Mixture Decreases Inspiratory Effort in Patients with Tracheal Stenosis. Respiration. 2019;97(1):42-51. doi: 10.1159/000492031. Epub 2018 Sep 18. PMID 30227423
- [Background] Guan WJ, Wei CH, Chen AL, Sun XC, Guo GY, Zou X, Shi JD, Lai PZ, Zheng ZG, Zhong NS. Hydrogen/oxygen mixed gas inhalation improves disease severity and dyspnea in patients with Coronavirus disease 2019 in a recent multicenter, open-label clinical trial. J Thorac Dis. 2020 Jun;12(6):3448-3452. doi: 10.21037/jtd-2020-057. No abstract available. PMID 32642277
- See also: WHO. Summary of probable SARS cases with onset of illness from 1 November 2002 to 31 July 2003. Dec 31, 2003. — https://www.who.int/csr/sars/country/table2004_04_21/en/
- See also: WHO. Middle East respiratory syndrome coronavirus (MERS-CoV). November, 2019. — http://www.who.int/emergencies/mers-cov/en/